CLINICAL TRIAL: NCT00878540
Title: Phase 1 Study of Mirtazapine in Healthy Subjects
Brief Title: Short-term Metabolic Effects of Mirtazapine in Healthy Subjects
Acronym: SMMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Prof. Florian Holsboer, Max-Planck-Institute of Psychiatry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: L2/2008; EudraCT-Nr.: 2008-002704-26
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: mirtazapine; metabolism; depression; Healthy males
MeSH Terms: conditions — Depression | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mirtazapine (Experimental)
  Interventions: Drug: mirtazapine

INTERVENTIONS:
Drug: mirtazapine — 30 mg mirtazapine once daily for 7 days
  Other Names: Remergil

SUMMARY:
The purpose of this study is to determine metabolic changes upon a 7 day medication of 30 mg mirtazapine per day in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 20-25 years
* Somatically and mentally healthy
* Normal body weight (body mass index (BMI)18.5-25)

Exclusion Criteria:

* Smoking within the last 6 months
* Medication within last 6 months
* Current or former psychiatric illness
* Positive family history (first grade relatives) for metabolic diseases
* Alcohol abuse
* Current or former illicit drug abuse
* Current or former drug abuse
* Known intolerance to, or former prescription of study medication
* Participation in other clinical trials at the same time or participation in clinical trials associated with administration of a drug within the last 6 months
* Homelessness
* Shift work within last 12 months
* Known hypersensitivity to mirtazapine or other components of the drug given
* Known epilepsy; glaucoma; liver, kidney, or heart disease; urinary dysfunction; hypotonia; diabetes or any other metabolic disease
* Known hematologic disease, especially agranulocytosis or leukopenia
* Blood donation within last 6 months prior to the begin of the study
* Hemoglobin below 13.5 mg/dL

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Metabolic changes upon a 7 day medication of 30 mg mirtazapine per day | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Florian Holsboer, MD, PhD, Principal Investigator — Max Planck Institute of Psychiatry, Munich
Locations (1):
- Max Planck Institue of Psychiatry, Munich, Germany

REFERENCES:
- [Derived] Lechner K, Heel S, Uhr M, Dose T, Holsboer F, Lucae S, Schaaf L, Fulda S, Kloiber S, Hennings JM. Weight-gain independent effect of mirtazapine on fasting plasma lipids in healthy men. Naunyn Schmiedebergs Arch Pharmacol. 2023 Sep;396(9):1999-2008. doi: 10.1007/s00210-023-02448-y. Epub 2023 Mar 9. PMID 36890393
- [Derived] Hennings JM, Heel S, Lechner K, Uhr M, Dose T, Schaaf L, Holsboer F, Lucae S, Fulda S, Kloiber S. Effect of mirtazapine on metabolism and energy substrate partitioning in healthy men. JCI Insight. 2019 Jan 10;4(1):e123786. doi: 10.1172/jci.insight.123786. PMID 30626746
- [Derived] Fulda S, Kloiber S, Dose T, Lucae S, Holsboer F, Schaaf L, Hennings J. Mirtazapine provokes periodic leg movements during sleep in young healthy men. Sleep. 2013 May 1;36(5):661-9. doi: 10.5665/sleep.2622. PMID 23633748